CLINICAL TRIAL: NCT06902168
Title: Effect of Diving and Aquatic Exercises on Muscle Spasticity and Motor Function in Children With Spastic Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Sarah Kotb Banawi, PhD in Philosophy, Faculty of Physical Education, Benha University, Egypt., Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC 4-2-2025
Record Dates: First submitted 2025-03-22; First posted 2025-03-30 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Diving; Aquatic; Muscle Spasticity; Motor Function; Children; Spastic Cerebral Palsy
MeSH Terms: conditions — Muscle Spasticity; Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intensive swimming program (Experimental): The participants will be enrolled in an intensive swimming program for 8 weeks (45 minutes) in the swimming pool. The swimming program will be to improve safety and functional independence in the water. The hydrotherapy will be performed at a swimming pool temperature suitable for the weather temperature.
  Interventions: Other: Intensive swimming program

INTERVENTIONS:
Other: Intensive swimming program — The participants will be enrolled in an intensive swimming program for 8 weeks (45 minutes) in the swimming pool. The swimming program will be to improve safety and functional independence in the water. The hydrotherapy will be performed at a swimming pool temperature suitable for the weather temperature.

SUMMARY:
This study aims to evaluate the effect of diving and aquatic exercises on muscle spasticity and motor function in children with spastic cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a common neurological disorders that affect movement and muscle coordination in childhood. Hydrotherapy is one of the most popular supplementary treatments for children with neuro-motor impairments, particularly children with CP.

Hydrotherapy may be more suitable for children with CP because of the properties of water, and it may be more motivating for children than land-based exercise. Buoyancy makes it easier for children with moderate to severe mobility limitations to move in the water than to move and exercise on land.

ELIGIBILITY:
Inclusion Criteria:

* Age from 2 to 5 years.
* Both sexes.
* Children diagnosed with spastic cerebral palsy, categorized according to the Gross motor function classification system (GMFCS) levels IV, V.

Exclusion Criteria:

* Botulinum toxin treatment or surgery in the preceding three months.
* Botox injections before or during the application of the program.
* Dorsal rhizotomy.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Estimated)
Dates: Start 2025-03-29 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Gross motor function measurement-66 | 8 weeks after intensive swimming program
  The gross motor function measurement-66 (GMFM-66) employs a four-point scoring system for each item. The 66 items are recorded according to the following classification: 0 = child unable to initiate the task; 1 = child initiates the task; 2 = child partially completes the task; 3 = child completes the task; and NT = not tested.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University (faculty of physical education), Banhā, Benha, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.